CLINICAL TRIAL: NCT06904625
Title: Comparison of Different Methods of CAPTure of Circulating Tumour Cells (CTC) in Patients With Metastatic Breast or Prostate Cancer
Acronym: CAPT CTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24GENE20
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer; Metastatic Prostate Cancer
Keywords: Circulating Tumor Cell; Metastatic Prostate Cancer; Metastatic Breast Cancer; CellSearch®; Parsortix®; SmartCatch®
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with metastatic breast cancer or prostate cancer (Other)
  Interventions: Other: Taking blood samples before starting treatment

INTERVENTIONS:
Other: Taking blood samples before starting treatment — For each patient included, a blood sample will be taken (37 mL in total) for the CTCs detection using the 3 techniques (CellSearch®, Parsortix® and SmartCatch®).
  For 3 patients only, an additional blood volume (18 mL) will also be collected for tcDNA detection (exploratory analysis of 3 patients).

SUMMARY:
This trial is a pilot, prospective, single-center study conducted in a population of patients with metastatic breast cancer (whatever the immunohistochemical subtype) or metastatic prostate cancer. The aim of this exploratory study is to compare the sensitivity of three different techniques (CellSearch®, Parsortix® and SmartCatch®) in detecting circulating tumor cells (CTCs). After the patient's agreement, and before starting anti-tumor treatment, a blood sample will be taken using the 3 different CTC detection techniques.

Each patient will participate in the study for one day.

A total of 36 evaluable patients (18 patients with metastatic breast cancer and 18 patients with metastatic prostate cancer) will be included in this interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with breast cancer (whatever the immunohistochemical subtype: triple-negative, RH+/HER2-negative or HER2-positive) or prostate cancer, multi-metastatic, eligible for a new line of treatment.
2. Patient not yet initiated on a new specific treatment for breast or prostate cancer at inclusion.
3. Age ≥ 18 years and WHO ≤ 2
4. Patient affiliated to Social Security scheme in France.
5. Patient having signed informed consent prior to inclusion in the study and prior to any study-specific procedures.

Exclusion Criteria:

1. Associated pathology(ies) likely to prevent the study procedure from running smoothly
2. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures stipulated in the study protocol.
3. Patient deprived of liberty or under legal protection (guardianship, legal protection)
4. Patient who has had another solid tumor (excluding carcinoma in situ of the breast or cervix) within 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with at least one additional CTC detected by the SmartCatch® method compared with the standard approach (CellSearch®). | 9 months after the study start
  It is defined by the ratio of the number of patients with at least one additional CTC detected by the SmartCatch® method compared with the standard approach (CellSearch®) to the total number of patients.

SECONDARY OUTCOMES:
The rate of patients with CTCs (CK+/CD45-) detected by each technique (CellSearch®, Parsortix® and SmartCatch®). | 9 months after the study start
  This is defined as the ratio of the number of patients with CTCs detected by the technique to the total number of patients.
The number of total CTCs (EpCAM+/CK+/CD45- and EpCAM-/CK+/CD45-) detected by the different techniques (CellSearch®, Parsortix® and SmartCatch®). | 9 months after the study start

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France